CLINICAL TRIAL: NCT06053515
Title: Rosie the Chatbot: Leveraging Automated and Personalized Health Information Communication to Reduce Disparities in Maternal and Child Health
Brief Title: Rosie the Chatbot: Leveraging Automated and Personalized Health Information Communication
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Maryland, College Park (Other)
Collaborators: National Institutes of Health (NIH) (NIH); National Institute on Minority Health and Health Disparities (NIMHD) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Supportive Care
Other Study IDs: 5R01MD016037-03 (NIH); 5R01MD016037-03 (NIH); 3R01MD016037-03S1 (NIH)
Record Dates: First submitted 2023-09-15; First posted 2023-09-25 (Actual); Last update posted 2024-04-17 (Actual); Status verified 2024-04

CONDITIONS: Pregnancy; Postpartum Depression; Infant Development; Infant Conditions
Keywords: chatbot; health information; racial/ethnic health disparities; maternal and child health; artificial intelligence; question-answering models
MeSH Terms: conditions — Depression, Postpartum

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Rosie the Chatbot Group (Experimental): Participants in the Rosie the Chatbot Group will be taking a pre-test health survey, mid-test health survey, and post-test health survey. In addition, they will be expected to actively use the chatbot app by asking questions related to maternal and infant health and selecting "thumbs up or thumbs down" to provide feedback for questions' response and using the features (video library, resources page, frequently asked questions (FAQ), and daily syllabus).
  Interventions: Behavioral: Rosie the Chatbot
- Book Club Group (No Intervention): Participants in the Book Club Group will be taking a pre-test health survey, mid-test health survey, and post-test health survey. In addition, they will receive a monthly children's book, which they are expected to read with baby if parenting or individually if pregnant.

INTERVENTIONS:
Behavioral: Rosie the Chatbot — Participants in the intervention group will be using the chatbot to ask questions related to the mom and baby's health, provide feedback "selecting thumbs up or thumbs down" on the questions' response, and use the features (video library, resources page, frequently asked questions (FAQ), and daily syllabus). In addition, participants will be taking a pre-test health survey, mid-test health survey, and post-test health survey.
  Arms: Rosie the Chatbot Group

SUMMARY:
Rosie the Chatbot is an educational chatbot that moms can have on their computers or cellphones and will work by moms typing in their questions about pregnancy, health, infant milestones, and other variety of health related topics and receiving back a response immediately. Rosie only provides information from verified sources such as children's hospitals, health organizations and government agencies. Rosie does not ask moms to provide any personal information on her or her child, her chat is completely confidential, it works in English and Spanish and will be free.

DETAILED DESCRIPTION:
This study will examine whether the use of a chatbot to impart health information to minority women during pregnancy and postpartum period improves health care seeking behavior and maternal and infant health outcomes. This study does not involve administration of an investigational intervention and therefore poses minimal risk to participants.

Aim 1: Develop technology for a "chatbot" that will provide health information support to vulnerable mothers the moment they need it.

Aim 2: Evaluate the use of Rosie on maternal and infant outcomes. Aim 3: Release an open-source packet for the construction of a chatbot.

* Participants in the study will be randomly assigned into one of two groups, Rosie the Chatbot group (treatment group) and Book Club group (control group).
* Participants in the Rosie the Chatbot Group will be taking a pre-test health survey, mid-test health survey, and post-test health survey. In addition, they will be expected to actively use the chatbot app by asking questions related to maternal and infant health and selecting "thumbs up or thumbs down" to provide feedback for questions' response and use the features (video library, resources page, frequently asked questions (FAQ), and daily syllabus).
* Participants in the Book Club Group will be taking a pre-test health survey, mid-test health survey, and post-test health survey. In addition, they will receive a monthly children's book, which they are expected to read with baby if parenting or individually if pregnant.

ELIGIBILITY:
Inclusion Criteria:

* Age 14 years and older
* Racial minority women
* Pregnant or has an infant < 6 months
* Must be able to read English or Spanish

Exclusion Criteria:

* Mother younger than 14 years of age at time of child's birth.
* Non-hispanic white

Ages: 14 Years to 99 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Gender Based: Yes — Female at birth
Enrollment: 400 (Estimated)
Dates: Start 2023-10-09 (Actual); Primary Completion 2026-01-01 (Estimated); Study Completion 2026-06-30 (Estimated)

PRIMARY OUTCOMES:
Maternal postpartum depression | 12 months post randomization
  The investigators will utilize the Patient Health Questionnaire (PHQ-9) Scale to measure maternal depression. This scale can range from 0 to 27, since each of the 9 items can be scored from 0 (not at all) to 3 (nearly every day). Higher scores indicate worse depression severity.
Number of emergency room visits | 12 months post randomization
  The investigators will measure the number of visits to the emergency room.
Attendance of well-baby visits (preventive healthcare visits) | 12 months post randomization
  The investigators will measure the number of well-baby visits.

CONTACTS AND LOCATIONS:
Overall Officials: Quynh C Nguyen, PhD, Principal Investigator — University of Maryland; Elizabeth M Aparicio, PhD, LCSW-C, Principal Investigator — University of Maryland
Locations (1):
- University of Maryland, College Park, Maryland, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Mane HY, Channell Doig A, Marin Gutierrez FX, Jasczynski M, Yue X, Srikanth NP, Mane S, Sun A, Moats RA, Patel P, He X, Boyd-Graber JL, Aparicio EM, Nguyen QC. Practical Guidance for the Development of Rosie, a Health Education Question-and-Answer Chatbot for New Mothers. J Public Health Manag Pract. 2023 Sep-Oct 01;29(5):663-670. doi: 10.1097/PHH.0000000000001781. PMID 37478093
- [Derived] Peters CJ, Aldana Lainez V, Clark K, Jasczynski M, Nguyen QC, Norell EM. Using an AI-powered Mobile Application Chatbot to Address Maternal Depression Indicators and Inquiries in the Perinatal and Postpartum Periods: A Multimethod Analysis. Inquiry. 2026 Jan-Dec;63:469580261417580. doi: 10.1177/00469580261417580. Epub 2026 Jan 29. PMID 41607314
- [Derived] Nguyen QC, Norell EM, Mane H, Yue X, Srikanth NP, Peters CJ, Gutierrez FXM, Kurella E, Dipankar P, Salazar D, Mullaputi PSP, Alibilli A, Santhosh A, He X, Boyd-Graber J, Nguyen TT. Developing an artificial intelligence-powered question-and-answer chatbot with English-Spanish capabilities for new mothers. JAMIA Open. 2026 Jan 6;9(1):ooaf169. doi: 10.1093/jamiaopen/ooaf169. eCollection 2026 Feb. PMID 41502532
- [Derived] Nguyen QC, Aparicio EM, Jasczynski M, Channell Doig A, Yue X, Mane H, Srikanth N, Gutierrez FXM, Delcid N, He X, Boyd-Graber J. Rosie, a Health Education Question-and-Answer Chatbot for New Mothers: Randomized Pilot Study. JMIR Form Res. 2024 Jan 12;8:e51361. doi: 10.2196/51361. PMID 38214963
- See also: Rosie aims to help close the racial gap in maternal and infant health disparities by providing new mothers with easy access to reliable health information. — https://www.ncbi.nlm.nih.gov/pmc/articles/PMC10372746/